CLINICAL TRIAL: NCT03586375
Title: Clinical and Cost Evaluation of Intensive Support Teams (IST) for Adults With Intellectual Disabilities and Challenging Behaviour
Brief Title: Intensive Support Teams Study
Acronym: IST-ID
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 16/0456
Record Dates: First submitted 2018-07-02; First posted 2018-07-13 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intensive Support Team Care — Intensive Support Teams (ISTs) are specialist teams which have been advocated for many years as the right services to help people with intellectual disabilities (ID) and challenging behaviour stay in their local communities. They may be staffed by one or more professions, e.g. psychology, nursing, psychiatry, and usually deliver interventions such as positive behaviour support and accept people with ID who are in a crisis when challenging behaviour emerges or provide support when a person is admitted to a local inpatient facility.

SUMMARY:
About 17% of people with ID living in the community have challenging behaviour such as aggression to others or property, self-injury or hyperactivity. There are concerns that adults with ID and challenging behaviour over-use medication, spend large periods of time in hospital, and miss out on living in the community. Hospital care is expensive, and costs are increasing. NHS England has produced draft guidance about Intensive Support Teams (ISTs) proposing that they should be part of all community ID services in England. However, there is currently very little evidence about how effective ISTs are. The people who pay for Health and Social Care services (commissioners) would like more information, and this project aims to provide this.

We propose to do a project over 36 months. It will be in two parts. First we will find out about how many, and what type of ISTs exist in England, by asking service managers about their service, their staff, and the work they do. With this information, we will identify different models of ISTs. Then we will look at several services in each model to compare how they work with people with ID and other local services. We will collect data twice over 9 months to see which model(s) work best. We will also carry out interviews with people who use ISTs, family and paid carers, and referrers to ISTs to find out about their experiences of these services, and how happy they are with them. Analysing and putting this data together will tell us about how effective each of the models are at reducing challenging behaviours, how much they cost, and which one service users, their families and people who work in other connected services prefer most.

We will tell people about our results at conferences and in academic and services journals. We will ask our group of involved service-users and family carers to guide us, and help us tell other people about the results. We have a team of clinicians and academics who are experts in all aspects of the research, e.g. statistics, ID, service evaluations, and in running ISTs. We will follow research rules and recommendations to make sure we carry out safe, ethical and rigorous research.

DETAILED DESCRIPTION:
Approximately 17% of adults with intellectual disabilities (ID also called learning disabilities in the UK; constitute about 1% of the population; living in the community present with serious challenging behaviour including aggression self-injury or other socially inappropriate behaviours. As many as 100,000 children and adults are estimated to be at risk of admission to inpatient care due to the presence of such behaviours if they are not successfully managed in the community. There are ongoing concerns that these individuals are subject to increased rates of hospitalisation, unnecessary long term use of psychotropic medication, poorer health, abuse and exclusion. Intensive Support Teams (ISTs) are specialist teams which have been advocated for many years as the right services to help people with intellectual disabilities (ID) and challenging behaviour stay in their local communities. They may be staffed by one or more professions, e.g. psychology, nursing, psychiatry, and usually deliver interventions such as positive behaviour support and accept people with ID who are in a crisis when challenging behaviour emerges or provide support when a person is admitted to a local inpatient facility. ISTs are recommended to provide high quality proactive and responsive care aimed at avoiding unnecessary admissions or reducing inpatient length of stay and supporting people in the community. However, there is little evidence to recommend a preferred IST model and there has not been any comprehensive attempt to describe IST outcomes. NHS Commissioners require clear information about what works in order to fund appropriate services. NG11 (8) reports the state of evidence thus: "It is widely recognised that locally accessible care settings could be beneficial and could reduce costs but there is no strong empirical evidence to support this".

Objectives: 1. To create a typology of IST currently operating in England; 2. To generate evidence on the effectiveness of different IST models which best support improved outcomes for adults with challenging behaviour; 3. To estimate the costs of different IST models and investigate cost effectiveness; 4. To understand how ISTs impact on the lives of adults with ID and challenging behaviour, their families and the local services; 5. To generate evidence to inform and support decision making on commissioning IST for adults with ID and challenging behaviour.

Methods: the proposed study has two phases: phase 1 (9 months) includes a national survey (England) of ISTs. Service managers of community ID teams (CIDT) will be approached to first identify whether they have such a service locally and then a piloted and refined survey will be carried out. Outputs will include mapping the distribution of ISTs, developing of IST models and a description of the key characteristics of these models. Phase 2 (27months) includes a mixed methods evaluation of up to 4 IST models. We will collect both patient level outcomes, e.g challenging behaviour, risk, hospitalisations, service use etc, at two assessment points (baseline and 9 months) and service level outcomes (referrer satisfaction, reach, referral numbers) over 9 months. Statistical analysis will compare outcomes across ISTs and identify which are most associated with positive outcomes (e.g. improvement in challenging behaviour). The costs of delivering the different models will be calculated and compared across all models. We shall collect qualitative data to understand the experiences and views of key stakeholders and the impact of the different models. We shall follow with a project report and a wide range of dissemination activities, e.g. publications, contacts with NHS England and policy makers, commissioners (CCGs), clinicians etc.

Main benefits: In line with NHS England (NHSE) guidance in managing people with ID locally and effectively, the proposed work will provide commissioners and clinicians with the evidence they need to deliver high quality care to an under-served population group. The project maps onto principles 7 and 8 of the plan outlined in Building the Right Support which describes the objectives of community ID services in England.

ELIGIBILITY:
Inclusion Criteria:

Service users - Eligible to receive support from IST service; mild to profound intellectual disability; aged 18 years and over/ Service - IST adheres to one of chosen models, has been operational for at least 12 months, there is commitment to fund it for the study duration and it can achieve sample size estimates.

Exclusion Criteria:

Service users - Primary clinical diagnosis of personality disorder of substance misuse; relapse in pre-existing mental disorder; decision taken by clinical team that a referral to the study would be inappropriate (e.g., there is an open complaint investigation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with mild to profound intellectual disability
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Challenging behaviour Aberrant Behaviour Checklist-Community version (ABC-C) | 0-9 months
  This is an established and internationally used carer administered measure of challenging behaviour.

SECONDARY OUTCOMES:
Carer reported Psychopathology Assessment for Adults with Developmental Disabilities checklist (PASADD Checklist) | 0-9 months
  Screen for mental disorder.
Threshold Assessment Grid (TAG) | 0-9 months
  Clinical risk
QoL-Q Schalock and Keith 1993 | 0-9 months
  Quality of Life
EQ 5D | 0-9 months
  Health-related Quality of Life
Client Service Receipt Inventory (CSRI) | 0-9 months
  Service Use

CONTACTS AND LOCATIONS:
Locations (16):
- United Kingdom (16):
  - Devon Partnership NHS Trust, Barnstaple
  - Cheshire and Wirral Partnership NHS Foundation Trust, Chester
  - Derbyshire Healthcare NHS Foundation Trust, Derby
  - London North West University Healthcare NHS Trust, Ealing
  - Care Plus Group, Grimsby
  - Hertfordshire Partnership University NHS Foundation Trust, Hatfield
  - Barnet, Enfield and Haringey Mental Health Trust, London
  - Nottinghamshire Healthcare NHS Foundation Trust, Nottingham
  - Midlands Partnership NHS Foundation Trust, Shrewsbury
  - Southern Health Foundation Trust, Southampton
  - Somerset Partnership NHS Foundation Trust, Taunton
  - Cornwall Partnership NHS Foundation Trust, Truro
  - Hounslow & Richmond Community Healthcare, Twickenham
  - East London NHS Foundation Trust, Whitechapel
  - Worcestershire Health and Care NHS Trust, Worcester
  - South West Yorkshire Partnership NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hassiotis A, Kouroupa A, Jones R, Morant N, Courtenay K, Hall I, Crossey V, Romeo R, Taggart L, Langdon P, Ratti V, Kirchner V, Lloyd-Evans B. Clinical and cost evaluation of intensive support team (IST) models for adults with intellectual disabilities who display challenging behaviour: a comparative cohort study protocol. BMJ Open. 2021 Mar 30;11(3):e043358. doi: 10.1136/bmjopen-2020-043358. PMID 33785489